CLINICAL TRIAL: NCT04852237
Title: Is the Lack of Prior Exposure to Sperm Antigens Associated With Worse Neonatal and Maternal Outcomes? A 10 Years Single-center Experience Comparing ICSI-TESE Pregnancies From ICSI Pregnancies
Brief Title: Is the Lack of Prior Exposure to Sperm Antigens Associated With Worse Neonatal and Maternal Outcomes?
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 1916
Record Dates: First submitted 2021-03-30; First posted 2021-04-21 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Obstructive Azoospermia; Obstetric Complication
Keywords: Neonatal outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnancies from ICSI-TESE cycles for obstructive azoospermia.: Pregnancies occurred between January 2010 and December 2019 at Humanitas Fertility Center after ICSI-TESE cycles for obstructive azoospermia.
- Pregnancies from ICSI cycles with ejaculated sperm.: Pregnancies occurred between January 2010 and December 2019 at Humanitas Fertility Center after ICSI cycles with ejaculated sperm.

SUMMARY:
The objective of this study is to determine if the lack of exposure to sperm antigens is associated with worse maternal and neonatal outcomes in pregnancies obtained after ICSI (intracytoplasmic sperm injection)-TESE (testicular sperm extraction) for obstructive azoospermia.

The primary outcomes that will be investigated include:

* Maternal outcomes: live birth rate (LBR), abortion rate, and the rate of the main obstetrics complication, such as pre-eclampsia, gestational hypertension and diabetes mellitus.
* Neonatal outcomes: gestational age, prematurity rate, birth weight, sex ratio, 1- and 5-min APGAR, birth defects.

DETAILED DESCRIPTION:
Several studies investigated the role of paternal factors in the development of preeclampsia; in particular, they analyzed the correlation between the vaginal exposure to male partner's semen and the incidence of preeclampsia, observing both a reduced risk of preeclampsia after prolonged exposure to the paternal seminal fluid and a higher incidence of preeclampsia in pregnancies conceived with a new father or with sperm donor. This leads to the hypothesis of an immunological role for sperm in inducing a mucosal immune tolerance-like status at the level of the uterus that could be critical in the subsequent implantation.

Previous studies also examined the neonatal outcomes from pregnancies obtained from surgically retrieved sperm, either epididymal or testicular sperm, and underlined that there is not overall increased risk in neonatal outcomes.

Our study aims at having a complete view on paternal, maternal and neonatal information and a follow up, that allows to correct possible confounders and to analyze a wider group of outcomes.

ELIGIBILITY:
Inclusion Criteria for case arm:

* primary infertility
* diagnosis of obstructive azoospermia
* ICSI-TESE cycles

Inclusion Criteria for control arm:

* primary infertility
* ICSI cycles with sperm from ejaculate

Exclusion Criteria:

* pre-gestational hypertension
* pre-gestational diabetes

Ages: 18 Years to 43 Years | Sex: All
Age Groups: Adult
Study Population: The study database will include all the pregnancies occurred between January 2010 and December 2019 at Humanitas Fertility Center after ICSI-TESE cycles for obstructive azoospermia.
  A comparison of maternal and neonatal outcomes will be performed among the above-mentioned pregnancies and pregnancies from ICSI cycles with ejaculated sperm of couples with different indications occurred in the same period of time.
  The controls will be matched to the cases for the principal risk factors for adverse maternal and neonatal outcomes (maternal age, BMI) with a ratio of 1:2.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Live birth rate (LBR) | 10 years
  Rate of delivery of a living baby after at least 22 weeks of gestation
Abortion Rate (AR) | 10 years
  Proportion of clinical pregnancies who failed to continue beyond 22 weeks of gestation
Maternal complications rate | 10 years
  Incidence of the obstetric complications, such as pre-eclampsia, gestational hypertension and diabetes, placenta previa and placental abruption.
Gestational age | 10 years
  Mean gestational age of the pregnancies considered (written with both weeks and days; eg, 39 weeks and 0 days)
Prematurity rate | 10 years
  Rate of pregnancies lasted less than 37 weeks and 0 days
Birth weight | 10 years
  Mean birth weight of the neonates, written in grams.
Sex ratio | 10 years
  Ratio between males and females among the newborns
1- and 5-min APGAR | 10 years
  Objective score of the condition of a baby after birth, at 1 and 5 minutes from the delivery (from 1 to 10 points).
Incidence of congenital defects | 10 years
  Incidence of congenital malformations, deformations and chromosomal abnormalities among the newborns of the study group (eg. clubfoot deformity, anorectal malformations, heart defects, ...)

REFERENCES:
- [Background] Robertson SA, Sharkey DJ. Seminal fluid and fertility in women. Fertil Steril. 2016 Sep 1;106(3):511-9. doi: 10.1016/j.fertnstert.2016.07.1101. Epub 2016 Jul 30. PMID 27485480
- [Background] Verwoerd GR, Hall DR, Grove D, Maritz JS, Odendaal HJ. Primipaternity and duration of exposure to sperm antigens as risk factors for pre-eclampsia. Int J Gynaecol Obstet. 2002 Aug;78(2):121-6. doi: 10.1016/s0020-7292(02)00130-3. PMID 12175712
- [Background] Wang JX, Knottnerus AM, Schuit G, Norman RJ, Chan A, Dekker GA. Surgically obtained sperm, and risk of gestational hypertension and pre-eclampsia. Lancet. 2002 Feb 23;359(9307):673-4. doi: 10.1016/S0140-6736(02)07804-2. PMID 11879865
- [Background] Di Mascio D, Saccone G, Bellussi F, Vitagliano A, Berghella V. Type of paternal sperm exposure before pregnancy and the risk of preeclampsia: A systematic review. Eur J Obstet Gynecol Reprod Biol. 2020 Aug;251:246-253. doi: 10.1016/j.ejogrb.2020.05.065. Epub 2020 Jun 1. PMID 32544753
- [Background] Dekker G, Robillard PY, Roberts C. The etiology of preeclampsia: the role of the father. J Reprod Immunol. 2011 May;89(2):126-32. doi: 10.1016/j.jri.2010.12.010. Epub 2011 May 6. PMID 21529966
- [Background] Andraweera P, Roberts CT, Leemaqz S, McCowan L, Myers J, Kenny LC, Walker J, Poston L, Dekker G; SCOPE Consortium. The duration of sexual relationship and its effects on adverse pregnancy outcomes. J Reprod Immunol. 2018 Aug;128:16-22. doi: 10.1016/j.jri.2018.05.007. Epub 2018 May 18. PMID 29803191
- [Background] Klonoff-Cohen HS, Savitz DA, Cefalo RC, McCann MF. An epidemiologic study of contraception and preeclampsia. JAMA. 1989 Dec 8;262(22):3143-7. PMID 2810672
- [Background] Robillard PY, Dekker G, Chaouat G, Hulsey TC, Saftlas A. Epidemiological studies on primipaternity and immunology in preeclampsia--a statement after twelve years of workshops. J Reprod Immunol. 2011 May;89(2):104-17. doi: 10.1016/j.jri.2011.02.003. Epub 2011 May 4. PMID 21543120
- [Background] Jin L, Li Z, Gu L, Huang B. Neonatal outcome of children born after ICSI with epididymal or testicular sperm: A 10-year study in China. Sci Rep. 2020 Mar 20;10(1):5145. doi: 10.1038/s41598-020-62102-y. PMID 32198466
- [Background] Belva F, De Schrijver F, Tournaye H, Liebaers I, Devroey P, Haentjens P, Bonduelle M. Neonatal outcome of 724 children born after ICSI using non-ejaculated sperm. Hum Reprod. 2011 Jul;26(7):1752-8. doi: 10.1093/humrep/der121. Epub 2011 Apr 21. PMID 21511713